CLINICAL TRIAL: NCT02478983
Title: A Randomized Comparison of LMA Supreme and LMA Proseal in Infants Below 10kg
Brief Title: A Randomized Comparison of LMA (Laryngeal Mask Airway) Supreme and LMA Proseal in Infants Below 10kg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Chaw Sook Hui, Dr., University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 995.7
Record Dates: First submitted 2015-06-07; First posted 2015-06-23 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Laryngeal Mask Airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LMA Supreme (Experimental): 1 arm will receive LMA supreme for airway management
  Interventions: Device: LMA Supreme
- LMA Proseal (Active Comparator): 1 arm will receive LMA Proseal for airway management
  Interventions: Device: LMA Proseal

INTERVENTIONS:
Device: LMA Supreme — The device will be inserted according to manufacturer's guideline. Time of insertion will be recorded. The oropharyngeal airway leak pressure will be measured when the device successfully inserted. The time taken to insert the LMA is recorded and the insertion success rate is documented. The larynx will be visualized with fibreoptic bronchoscope inserted through the LMA. Intraoperative complications will be recorded.
  Arms: LMA Supreme
Device: LMA Proseal — The device will be inserted according to manufacturer's guideline. Time of insertion will be recorded. The oropharyngeal airway leak pressure will be measured when the device successfully inserted. The time taken to insert the LMA is recorded and the insertion success rate is documented. The larynx will be visualized with fibreoptic bronchoscope inserted through the LMA. Intraoperative complications will be recorded.
  Arms: LMA Proseal

SUMMARY:
The investigators conduct this study to evaluate the clinical efficacy of size 1 and 1.5 supreme LMA compared to proseal LMA for infants weighing <10kg.

DETAILED DESCRIPTION:
This is a randomized prospective study to compare the clinical efficacy and safety for size 1 and 1.5 LMA supreme and LMA Proseal. The airway leak pressure of these 2 devices will be compared and other parameters such as time to insertion, insertion success rate, fibreoptic glottic view and intraoperative complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Weight of < 10kg
* ASA (American Society of Anesthesiologists) I-II
* Infants undergoing elective surgery under general anaesthesia using supraglottic airway device.
* Informed consent obtained from parents.

Exclusion Criteria:

* ASA III-IV and emergency surgery
* Neonates and ex-premature babies with post conceptual age <55 weeks.
* Infants with history of difficult airway.
* Infants with features of difficult intubation.
* Active upper respiratory tract infection
* Infants with pulmonary disease
* Infants with history of gastroesophageal reflux disease
* Infants with risks of regurgitation and aspiration.

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | intraoperative
  The measurement of oropharyngeal airway pressure when airway leak occurred

SECONDARY OUTCOMES:
Insertion success rate | intraoperative
  The number of attempts for successful placement of the supraglottic airway is recorded.
Fibreoptic glottis view | intraoperative
  Fibreoptic glottis view will be recorded according to a grading system
Intraoperative complications | intraoperative
  Complications such as loss of airway patency, desaturation, regurgitation of gastric contents, laryngospasm, bronchospasm and airway trauma will be recorded
Time to insertion | intraoperative
  Time from picking up the supraglottic airway device to the first detection of capnography square wave

CONTACTS AND LOCATIONS:
Overall Officials: Sook Hui Chaw, M.Med, Principal Investigator — University of Malaya
Locations (1):
- Faculty of Medicine, University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No